CLINICAL TRIAL: NCT01092273
Title: Bimatoprost Versus Travoprost in an Egyptian Population: A Hospital-Based Prospective Randomized Study.
Brief Title: Bimatoprost Versus Travoprost at Cairo University
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Other Study IDs: Prostaglandins-Cairo-1A
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2008-01

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma and Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bimatoprost versus Travoprost

SUMMARY:
Bimatoprost has been shown to provide effective IOP lowering in patients of all races. Conversely, travoprost has been shown to be more effective in black patients than in Caucasians in some studies. However, Noecker et al 2004 compared bimatoprost with travoprost in African-Americans with glaucoma or OHT, and found that bimatoprost was more likely than travoprost to achieve target pressure at 3 months.

These racial differences in efficacy of these medications warrant further investigations. The investigators study aim to compare the IOP-lowering efficacies of bimatoprost and travoprost in an Egyptian population with primary open-angle glaucoma (OAG) or ocular hypertension (OHT).

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma and Ocular Hypertension

Exclusion Criteria:

* Any ocular disease or medication that may raise the intraocular pressure.

Ages: 20 Years to 72 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospital Based Study at Cairo University and Al Nour Eye Hospital
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
Percentage of intraocular pressure lowering of bimatoprost versus travoprost.

SECONDARY OUTCOMES:
Rate of development of complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/19726422